CLINICAL TRIAL: NCT02395302
Title: Evaluation of a Dual Action Pneumatic Compression Device: Patient Ease of Use and Comfort in Patients With Venous Leg Ulcers
Brief Title: Evaluation of a Dual Action Pneumatic Compression System: Tolerance and Comfort in Patients With Venous Leg Ulcers (VLUs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6020
Record Dates: First submitted 2015-03-10; First posted 2015-03-23 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Venous Leg Ulcer; Chronic Venous Insufficiency; Venous Stasis Ulcer; Venous Ulcer; Venous Insufficiency
MeSH Terms: conditions — Varicose Ulcer; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dual Action Pneumatic Compression (Experimental): Dual action pneumatic compression device that provides both sustained compression while ambulatory, and intermittent pneumatic compression when connected to an alternating current (AC) outlet.
  Interventions: Device: Dual Action Pneumatic Compression

INTERVENTIONS:
Device: Dual Action Pneumatic Compression — Wear in sustained mode for 14 hours and pneumatic compression mode for 3 hours during the 4 week treatment period.
  Other Names: ACTitouch system

SUMMARY:
The purpose of the study is to assess treatment tolerance and comfort in chronic VLUs after 4 weeks of treatment using a dual action pneumatic compression device.

DETAILED DESCRIPTION:
Subjects with a chronic venous leg ulcer will participate in a 2 week run in phase using standard of care multi-layer bandaging before receiving 4 weeks of treatment using a pneumatic compression device. Subjects will be seen in clinic weekly for an evaluation, complete symptom and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age or legal age at the time of enrollment.
* Chronic venous insufficiency confirmed by ultrasound within previous 12 months.
* Active ulceration (CEAP classification of C6)
* Ulcer duration: ≥ 2 month but not greater than 24 months - non healing VLU with conservative treatment.
* Ulcer size ≥ 2cm2 ≤ 50cm2
* Leg circumferences within the following range:Ankle - 12 to 44cm;Calf - 22 to 60cm; Below knee - 22 to 68cm

Exclusion Criteria:

* Target ulcer or any other ulcer on the study limb involves exposure of tendon, muscle, or bone.
* Greater than 3 separate full thickness ulcers on the study limb
* Target ulcer is of non-venous etiology (sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma, malignancy).
* Treatment of the target ulcer with living cellular therapy within 30 days of the time of enrollment.
* History of an acute deep vein thrombosis (DVT) or pulmonary embolism (PE) within the last 3 months.
* Either the dorsalis pedis (DP) or posterior tibial (PT) systolic pressure < 80mmHg for diabetic patients or < 60mmHg for non-diabetic patients on study limb or transcutaneous partial pressure oxygen (Tcp02) ≤ 30mmHg or great toe systolic pressure ≤ 40mmHg.
* Acute thrombophlebitis.
* History of pulmonary edema or decompensated congestive heart failure.
* Currently has an active infection of the skin such as cellulitis requiring antibiotics.
* History of cancer within the last 5 years with the exception of treated non-melanoma skin cancer or cervical carcinoma in situ.
* Poorly controlled diabetes with a Hemoglobin A1c (HbA1c) value of >12%.
* Changes to medications that affect edema within the last 30 days
* Need for current and ongoing therapy with corticosteroids (exception for continued low dose usage) or cytotoxic drugs or the current use of Daflon 500.
* Currently pregnant or trying to become pregnant.
* Inability or unwillingness to participate in all aspects of study protocol.
* Currently participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Marston, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (6):
- United States (6):
  - Center for Clinical Research, San Francisco, California
  - University of Miami School Hospital, Miami, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - St. Luke's Roosevelt Hospital Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dual Action Pneumatic Compression: Dual action pneumatic compression device that provides both sustained compression while ambulatory, and intermittent pneumatic compression when connected to an alternating current (AC) outlet. Subjects that received the dual action pneumatic compression device were instructed to use the device in sustained mode for fourteen hours per day and in intermittent mode for three hours per day during the four week treatment period.
Period: Overall Study
Arm/Group | Dual Action Pneumatic Compression
Started | 28
Completed | 14
Not Completed | 14
Not completed — Screen Failure | 3
Not completed — Run In Failure | 7
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Demographic information for 27 of the 28 study subjects was collected. One study subject was withdrawn from the study before demographic information was collected.
Groups:
- Dual Action Pneumatic Compression: Dual action pneumatic compression device that provides both sustained compression while ambulatory, and intermittent pneumatic compression when connected to an AC outlet.
  Dual Action Pneumatic Compression: Wear in sustained mode for 14 hours and pneumatic compression mode for 3 hours during the 4 week treatment period.
Arm/Group | Dual Action Pneumatic Compression
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Agreed With Tolerance and Comfort Questionnaire Items After Using a Dual Action Pneumatic Compression Device
Description: A questionnaire that was completed after receiving four weeks of treatment from a dual action pneumatic compression device. Questions listed below:
  1. The device was comfortable to wear during Sustained Compression Mode.
  2. The device was comfortable to wear during Intermittent Compression Mode.
  3. The noise from the device was not bothersome.
  4. The device was easy to put on.
  5. The device was easy to take off.
  6. The device was easy to use.
  7. The device was light-weight and portable.
  8. The use of the device helped my wound heal faster.
  9. I would use the device again on another wound in the future.
  10. Since using the device, my quality of sleep has improved.
  11. It was a burden to come to the wound care clinic for my dressing changes.
  12. The use of the device did not restrict many of my normal activities.
  13. The device was cumbersome and interfered with my mobility.
  14. I was able to work while being treated with the device.
Time Frame: 4 weeks
Population: The Tolerance and Comfort questionnaire was completed at study exit by 16 participants (13 of the 16 total subjects completed the study, 2 were withdrawn by their site's Investigator, and 1 voluntarily withdrew).
  Six participants were not employed during the time of questionnaire completion. Question 14 was not applicable to these participants.
Measure: Count of Participants; unit: Participants
Groups:
- Dual Action Pneumatic Compression: Dual action pneumatic compression device that provides both sustained compression while ambulatory, and intermittent pneumatic compression when connected to an AC outlet.
Arm/Group | Dual Action Pneumatic Compression
Number analyzed (Participants) | 16
Participants
  Participants who agreed with Question 1 | 12
  Participants who agreed with Question 2 | 8
  Participants who agreed with Question 3 | 9
  Participants who agreed with Question 4 | 15
  Participants who agreed with Question 5 | 15
  Participants who agreed with Question 6 | 15
  Participants who agreed with Question 7 | 11
  Participants who agreed with Question 8 | 8
  Participants who agreed with Question 9 | 13
  Participants who agreed with Question 10 | 7
  Participants who agreed with Question 11 | 6
  Participants who agreed with Question 12 | 9
  Participants who agreed with Question 13 | 9
  Participants who agreed with Question 14: number analyzed (Participants) | 10
  Participants who agreed with Question 14 | 8

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Dual Action Pneumatic Compression
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 10/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Action Pneumatic Compression (N=28)
Pain in extremity (Injury, poisoning and procedural complications) | 3 (4)
Blister (Skin and subcutaneous tissue disorders) | 3 (3)
Migraine (General disorders) | 1 (2)
Skin ulcer (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Application site erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Cramping (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less